CLINICAL TRIAL: NCT01445379
Title: A Phase I Study of Ipilimumab (Anti-CTLA-4) in Children, Adolescents, and Young Adults With Treatment Refractory Cancer
Brief Title: Phase I Study of Ipilimumab (Anti-CTLA-4) in Children and Adolescents With Treatment-Resistant Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 080007; 08-C-0007; NCT00556881 (obsolete NCT alias)
Record Dates: First submitted 2011-09-30; First posted 2011-10-03 (Estimated); Last update posted 2019-12-17 (Actual); Status verified 2015-11-13

CONDITIONS: Sarcoma; Wilm's Tumor; Lymphoma; Neuroblastoma
Keywords: Solid Tumor; Monoclonal Antibody; Pediatrics; Pharmacokinetics; Immunotherapy; Sarcoma; Lymphoma; Neuroblastoma
MeSH Terms: conditions — Sarcoma; Wilms Tumor; Lymphoma; Neuroblastoma | interventions — Ipilimumab

ARMS (1):
- 1 (Experimental): Ipilumumab (DSE) given on day 1 of 21 day cycle for 4 cycles, from cycle 5+ ipilumumab will be given ~every 12wks
  Interventions: Drug: Ipilimumab

INTERVENTIONS:
Drug: Ipilimumab — Dose Level Escalation: 1mg/kg, 3mg/kg, 5mg/kg, 10mg/kg

SUMMARY:
This study will examine the safety and efficacy of ipilimumab-an experimental cancer treatment drug used to boost immune response-in children, adolescents, and young adults. Ipilimumab may allow immune cells to react to and destroy abnormal cells in the body, and has been tested in adults for a variety of cancers and has shown responses in some research studies. Because ipilimumab has not been tested in children, adolescents, or young adults, it is considered an experimental drug. The purposes of this research study are to determine the highest safe dose of ipilimumab for children, adolescents, and young adults with solid tumor cancers; examine its effectiveness and possible side effects; and better understand how the body and the immune system process it over time.

Candidates must be between 2 and 21 years of age and must have solid malignant tumors that have been resistant to standard therapy. Volunteers will be screened with a medical history, a clinical examination, and computerized scans such as magnetic resonance imaging (MRI). Participants must have completed their last dose of chemotherapy, radiation, chemotherapy, or antibody or investigational therapy at least four weeks prior to enrollment.

During the study, participants will receive an intravenous dose of ipilimumab once every three weeks. The infusion of ipilimumab will last 90 minutes, and the participant s vital signs will be monitored while the medicine is infusing and several times in the first 24 hours after the first dose (requiring a hospital stay during that time). If the participant is able to tolerate the first dose of ipilimumab, further doses (called cycles ) may be received on an outpatient basis. Blood and urine tests will be given on a regular basis during these cycles. After four cycles, participants whose tumors do not grow and who do not have unacceptable side effects will continue to receive ipilimumab every three months to maintain the current condition, until researchers conclude the study.

DETAILED DESCRIPTION:
Background:

Solid tumors represent approximately one fourth of cancer diagnoses in children. Despite intensive regimens, patients with metastatic or recurrent solid tumors have unsatisfactory survival rates. Therefore new therapies are needed to improve outcomes.

Accumulating preclinical and clinical evidence supports the use of biologic approaches to heighten antitumor immunity in order to improve the effectiveness of immune based therapy. Both directly activating immune based therapies such as cytokines and tumor vaccines as well as therapies which disrupt negative counterregulatory signals such as those mediated by CTLA-4:B7 may enhance existent antitumor immune responses.

Antibodies directed against CTLA-4 potently augment immune responses in animal models and anti-CTLA-4 antibodies have demonstrated antitumor effects in a variety of preclinical tumor models.

Phase I and phase II studies using ipilimumab have been performed in adults with a variety of tumor types. Clinical responses have been observed in renal cell carcinoma, melanoma, and prostate cancer. No trials have yet been performed to evaluate ipilimumab in children with malignancy.

Objectives:

To determine the tolerance and toxicity profile of ipilimumab at a range of doses up to, but not exceeding, the highest dose tolerated in adults, in patients less than or equal to 21 years of age with refractory solid tumors.

To assess the pharmacokinetics of ipilimumab administered intravenously in patients less than or equal to 21 years of age with advanced and/or refractory solid tumors.

Eligibility:

Patients must be 1-21 years of age at the time of enrollment with solid malignant tumors refractory to standard therapy.

Design:

A Phase I dose finding study with 4 planned dose levels.

Three patients will be enrolled at each dose level with an expanded cohort of 12 at the highest or maximum torlerated dose with intent to include 6 patients < 12 years.

Re-induction with 4 infusions of ipilimumab at the assigned dose followed by another maintenance phase is possible for subjects who have progressed during maintenance therapy.

ELIGIBILITY:
* INCLUSION CRITERIA:

AGE: Patients must be greater than or equal to 1 years and less than or equal to 21 years of age.

DIAGNOSIS: Histologically confirmed solid tumors, which may include but are not limited to rhabdomyosarcoma and other soft tissue sarcomas, Ewing s sarcoma family of tumors, osteosarcoma, neuroblastoma, Wilm s tumor, Hodgkin's or non-Hodgkin's lymphoma. Patients with melanoma are eligible. Patients with a previous history of CNS metastases are eligible if the metastases have been treated with surgery and/or radiotherapy, are clinically stable as evidenced by no requirements for corticosteroids, the patient has no evolving neurologic deficits and no progression in residual brain abnormalities without specific therapy over 4 weeks.

MEASURABLE/EVALUABLE DISEASE: Patients must have measurable or evaluable tumors.

PRIOR THERAPY:

* The patient s cancer must have relapsed following or failed to respond to standard therapy and/or the patient s current disease state must be one for which there is no known curative therapy or therapy proven to prolong survival.
* Patients must have completed their last dose of irradiation, chemotherapy, monoclonal antibody, or investigational therapy at least 4 weeks prior to enrollment. For patients who have undergone autologous stem cell transplantation, at least 3 months must have elapsed since transplant.
* Patients must have recovered from the toxic effects (to a grade 1 or less) of all prior therapy prior to enrollment, with the exception of the following:

  * Hematological toxicity: recovery to levels required below
  * Low electrolyte levels (Such individuals should receive appropriate supplementation)
  * For patients on anticoagulant therapy or with pre-existing coagulation abnormalities, PT, PTT must return to baseline.
  * Liver function tests must resolve to values required below
  * Grade 3 hypoalbuminemia
  * Alopecia
  * Sterility

PERFORMANCE STATUS: Patients greater than 10 years old must have a Karnofsky Score of greater than or equal to 50 and children less than 10 years old must have a Lansky score of greater than 50. Patients who are unable to walk because of paralysis or weakness, but who are up in a wheelchair will be considered ambulatory for the purpose of calculating the performance score.

HEMATOLOGIC FUNCTION: Patients must have adequate bone marrow function, defined as a peripheral absolute granulocyte count of greater than or equal to 1000/microL, hemoglobin greater than or equal to 8 gm/dl, and a platelet count greater than or equal to 50,000/microL (may be corrected with transfusions).

HEPATIC FUNCTION: Aspartate transaminase (AST) and alanine transaminase (ALT), less than or equal to 2.5-fold the upper limit of normal (ULN). Normal total bilirubin.

RENAL FUNCTION: Patients must have normal age-adjusted serum creatinine (see table below) OR a creatinine clearance greater than or equal to 70 mL/min/1.73 m(2).

MAXIMUM SERUM CREATININE LEVEL FOR AGE:

* For children whose age is less than or equal to 5 years, 0.8 mg/dL
* For children whose age is greater than 5 but less than or equal to 10, 1.0 mg/dL
* For children whose age is greater than 10 but less than or equal to 15, 1.2 mg/dL
* For children whose age is greater than 15, 1.5 mg/dL

INFECTIOUS DISEASE:

-A patient with viral hepatitis (HBV, HCV) or human immunodeficiency virus (HIV) will be excluded from trial to limit confounding variables in the assessment of the potential hepatic toxicity of ipilimumab and uncertain impact of ipilimumab administration on viral replication. Serology will not be required unless infection is clinically suspected. A positive hepatitis B titer does not exclude a patient if immunization has been performed and if there is no history of disease.

INFORMED CONSENT: All patients or their legal guardians (if the patient is less than 18 years old) must sign a document of informed consent (Pediatric Oncology Branch, NCI screening protocol for NIH patients) prior to performing studies to determine patient eligibility. After confirmation of eligibility, all patients or their legal guardians must voluntarily sign the IRB approved protocol specific informed consent to document their understanding of the investigational nature, the risks of this study and their willingness to receive the therapy and undergo the research studies involved including pharmacokinetic studies. The consent must be signed before any protocol related studies are performed (This does not include routine laboratory tests or imaging studies required to establish eligibility). When appropriate, pediatric patients will be included in all discussions in order to obtain verbal assent.

DURABLE POWER OF ATTORNEY (DPA): Patients who are greater than or equal to 18 years of age will be offered the opportunity to assign a DPA so that another person can make decisions about their medical care if they become incapacitated or cognitively impaired.

BIRTH CONTROL: Patients of childbearing or child-fathering potential must be willing to use a medically acceptable form of birth control which includes abstinence, while they are being treated on this study and for 60 days following the last dose. Females of childbearing potential must have a negative pregnancy test within 14 days prior to initiation of study therapy and prior to each additional dose of ipilimumab.

EXCLUSION CRITERIA:

* Primary brain tumors
* Clinically significant unrelated systemic illness, such as serious infections or organ dysfunction, which in the judgment of the Principal or Associate Investigators would compromise the patient s ability to tolerate the agents in this trial or are likely to interfere with the study procedures or results. This includes but is not limited to:

  * Critically-ill or medically unstable patients
  * Patients with active infection or other significant systemic illness
  * Patients with active diarrhea
  * Patients with active eye inflammation, uveitis
  * Presence of a symptomatic pleural effusion
  * Patients with symptoms of congestive heart failure or uncontrolled cardiac rhythm disturbance
  * History of malignant hyperthermia
  * Concurrent or history of autoimmune disease excluding stable asthma
  * Positive direct Coombs testing or history of hemolytic anemia
  * Patients with a history of ongoing or intermittent bowel obstruction
* Concurrent radiation
* Patients with a history of allogeneic bone marrow transplantation.
* Untreated CNS metastases will render the patient ineligible however patients with a previous history of CNS metastases are eligible if: the metastases have been treated with surgery and/or radiotherapy, are clinically stable as evidenced by no requirements for corticosteroids, the patient has no evolving neurologic deficits and no progression in residual brain abnormalities without specific therapy are eligible one week post radiation or radiosurgery. Patients with asymptomatic subcentemeric CNS lesions will be eligible for trial if no immediate radiation or surgery.
* Patients with a history of previous therapy with ipilimumab will be excluded from study participation.
* Treatment with any of the following immunomodulatory agents within 14 days prior to study entry:

  --Systemic corticosteroid therapy

  ---Erythropoeitin
* Retinoic acid

  * Fenretinide
  * Interferons or interleukins
  * Cytokine-fusion proteins
  * Growth hormone
  * IVIG
* Treatment with myeloid growth factors (GM-CSF or G-CSF) within 72 hours prior to study entry.
* Patients with autoimmune disease, including autoimmune hemolytic anemia, ulcerative and hemorrhagic colitis, endocrine disorders (e.g., thyroiditis, hyperthyroidism, hypothyroidism, autoimmune hypophysitis/hypopituitarism, and adrenal insufficiency),

sarcoid granuloma, myasthenia gravis, polymyositis, and Guillain-Barre syndrome.

* Pregnant or breastfeeding females are excluded because ipilimumab may be harmful to the developing fetus or nursing child.
* Concurrent administration of any other investigational agent.

Ages: 3 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 33 (Actual)
Dates: Start 2007-10-01; Primary Completion 2014-04-18 (Actual); Study Completion 2015-11-13 (Actual)

PRIMARY OUTCOMES:
To determine the tolerance and toxicity profile | 1 year
Pharmacokinetics | 1 year

SECONDARY OUTCOMES:
Evaluate immunomodulatory activity. | 2 years
Quantify antitumor effects | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Melinda S Merchant, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (3):
- United States (3):
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Memorial Sloan Kettering Cancer Center, New York, New York

REFERENCES:
- [Background] Linet MS, Ries LA, Smith MA, Tarone RE, Devesa SS. Cancer surveillance series: recent trends in childhood cancer incidence and mortality in the United States. J Natl Cancer Inst. 1999 Jun 16;91(12):1051-8. doi: 10.1093/jnci/91.12.1051. PMID 10379968
- [Background] Dunn GP, Old LJ, Schreiber RD. The three Es of cancer immunoediting. Annu Rev Immunol. 2004;22:329-60. doi: 10.1146/annurev.immunol.22.012703.104803. PMID 15032581
- [Background] Zou W. Immunosuppressive networks in the tumour environment and their therapeutic relevance. Nat Rev Cancer. 2005 Apr;5(4):263-74. doi: 10.1038/nrc1586. PMID 15776005